CLINICAL TRIAL: NCT06844097
Title: Testing the Effectiveness of an Intervention to Foster Cervical Cancer Screening Promotion for Latinx Trans Men Among Medical Students
Brief Title: Intervention for Medical Student to Promote Cervical Cancer Screening Among Latinx Transmasculine Individuals
Acronym: CC-Trained
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ponce Medical School Foundation, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2308159535R001; 2U54CA163071-11 (NIH)
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Clinical Competence; Medical Education; Cervical Cancer Screening
Keywords: Latinx transmaculine; Latinx Non-Binary; Medical Students; SGM Cancer Research; Efficacy Study; Cervical Cancer Prevention Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cervical Cancer Trans Inclusive Education (CC-TRAINED) Module (Experimental): Participants assigned to the experimental condition will receive the CC-TRAINED intervention.
  Interventions: Behavioral: Cervical Cancer Trans Inclusive Education (CC-TRAINED) Module
- Disaster Preparedness Course (Other): Participants randomized to the control condition will receive a Disaster Preparedness Course, addressing the basics of natural disaster preparedness
  Interventions: Behavioral: Disaster Preparedness Course

INTERVENTIONS:
Behavioral: Cervical Cancer Trans Inclusive Education (CC-TRAINED) Module — An online course designed to increase cervical cancer prevention clinical skills among medical students when working with Latinx transmasculine populations.
  Arms: Cervical Cancer Trans Inclusive Education (CC-TRAINED) Module
Behavioral: Disaster Preparedness Course — An online course designed to improve professionals' skills and competencies for engaging in disaster preparedness.
  Arms: Disaster Preparedness Course

SUMMARY:
The team aims to test the effectiveness of an intervention to increase gender-affirming cervical cancer prevention behaviors targeted at medical students studying in Puerto Rico and Florida. The team expects that after exposure to the intervention, relative to the control group, participants in the experimental condition will manifest more favorable changes in knowledge, attitudes, and behaviors of adequate care towards Latinx transmasculine and non-binary people.

DETAILED DESCRIPTION:
Transmen (TM) and non-binary individuals (NB; individuals assigned female sex at birth who identify as a man, male, or another diverse non-binary gender identity on the masculine spectrum) are at higher risk of screening-detectable cancers. Latinx TM-NB (LTM-NB) are at a higher risk for cervical cancer (CC) as they intersect two health disparity populations with high risk for this type of cancer (gender identity and ethnic minorities). Despite CC being highly preventable, LTM-NB individuals have been found to have lower rates of CC screening than cisgender female patients (persons who are not transgender). Unfortunately, findings from the team's previous funded studies with LTM-NB individuals in Puerto Rico (PR) and Florida evidence that providers lack knowledge regarding LTM-NB individual's healthcare needs, have negative stigmatizing attitudes, and manifest discriminatory behaviors in clinical interactions with LTM-NB individuals; which greatly limits their ability for engaging in recommended education and prevention guidelines of care for CC screening and prevention. In light of this, the research team (community stakeholders from PR and Mainland US, researchers, and providers) has developed a brief online intervention to improve medical students' competencies for cervical cancer education and screening promotion among LTM-NB individuals.

The proposed study aims to: 1) Test the effectiveness of the intervention in increasing medical students' knowledge, attitudes, and skills for providing healthcare to LTM-NB. , 2) Determine the acceptability, appropriateness, and feasibility of implementing the interventions in real-world medical educational settings.

While the team has preliminary data regarding the efficacy of the intervention, this pilot is proposing a rigorous study design: Aim 1 will measure the magnitude of effect of the intervention, and Aim 2 measures the implementation. This study will address cervical cancer disparities among LTM-NB individuals. The impact of this study will reveal new effective interventions and implementation strategies. The translational implications of this work will result in providing medical schools with a cross-cultural tool to train students on cervical cancer prevention for LTM-NB individuals.

ELIGIBILITY:
Inclusion Criteria:

* Medical student currently in third year of medical school training

Exclusion Criteria:

* Do not speak English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-07 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change cervical cancer preventive behaviors, as determined by the Cervical Cancer Preventive Behaviors Inventory | Baseline, immediately after the intervention
  The CCPBI includes 46 non-verbal and verbal behaviors that can be manifested during the SPS interactions with LTM. The team expects that following intervention exposure, relative to control group participants, intervention participants will manifest a higher mean number of CC preventive behaviors on the CCPBI outcome.
Change in LTMNB knowledge, as determined by Transmasculine knowledge index | Baseline, immediately after the intervention
  This measure assesses health professionals' knowledge of TM-specific health issues. Intervention participants, relative to controls, will have a higher mean knowledge (literacy) level regarding LTM issues.
Change negative attitudes towards LTMNB, as determined by the transgender stigma scale | Baseline, immediately after the intervention
  This scale measures stigma related to transgender identity among healthcare providers. Intervention participants, relative to controls, will have a lower mean level of stigmatizing attitudes toward LTM
Change negative and increase positive emotions related to LTMNB, as determined by the Emotional Reactions Scale | Baseline, immediately after the intervention
  This scale measures emotional reactions to LTMNB. Intervention participants, relative to control participants, will have an increase in the mean of positive emotions, and a reduction in the mean level of negative emotions.
Change cultural humility, as determined by the cross-cultural scale | Baseline, immediately after the intervention
  This adaptation of the Cross-Cultural Care Scale55 measures cultural humility preparedness and skills towards multiple identities. Intervention participants, relative to control participants, will have an increase in the mean of cultural humility.

SECONDARY OUTCOMES:
Sex as a biological variable | Baseline, immediately after the intervention
  Following NIH guidance regarding investigating differential effects of sex and gender, we will repeat all analyses twice, stratified by a) sex at birth and b) current gender identification, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Alixida Ramos Pibernus, PhD, Principal Investigator — Ponce Health Sciences University; Matthew B Schabath, PhD, Principal Investigator — H. Lee Moffit Cancer Center and Research Institute

IPD SHARING:
Plan to Share IPD: No